CLINICAL TRIAL: NCT05330949
Title: Retinal Microvascular Changes by Optical Coherence Tomography Angiography Compared to Maternal Uterine Artry Doppler in Screening for Hypertensive Disorders in High-risk Pregnancies
Brief Title: Optical Coherence Tomography Angiography Compared to Maternal Doppler in Screening for Hypertension in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Esmail Khalil Esmail, lecturer of Ophthalmology, Minia University
Other Study IDs: 294-2022
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Pregnancy Induced Hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- case group
  Interventions: Diagnostic Test: Optical coherence Tomography Angiography, Uterine artry doppler
- control
  Interventions: Diagnostic Test: Optical coherence Tomography Angiography, Uterine artry doppler

INTERVENTIONS:
Diagnostic Test: Optical coherence Tomography Angiography, Uterine artry doppler — vascular changes in retina by OCT angiography and uterine artry doppler in the first and second trimesters

SUMMARY:
Pregnancy related hypertension is one of the most prevalent obstetric complications. The aim of the study is to evaluate the validity and sensitivity of OCT angiography in prediction of pregnancy induced hypertensive disorders in comparison to maternal doppler in the first and second trimesters of pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the first and second trimesters

Exclusion Criteria:

* pregnant females with associated systemic vascular disease as diabetes, SLE

Ages: 22 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnant females
Study Population: two groups according to the risk of developing hypertension during pregnancy
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
validity and sensitivity of OCT angiography | 6 months
  sensitivity of OCTA in comparison to doppler in prediction of pregnancy related hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Minia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided